CLINICAL TRIAL: NCT01218867
Title: Phase I/II Study of Metastatic Cancer Using Lymphodepleting Conditioning Followed by Infusion of Anti-VEGFR2 Gene Engineered CD8+ Lymphocytes
Brief Title: CAR T Cell Receptor Immunotherapy Targeting VEGFR2 for Patients With Metastatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No objective responses were observed.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110013; 11-C-0013
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Cancer; Metastatic Melanoma; Renal Cancer
Keywords: Clinical Response; Metastatic Cancer; Immunotherapy; Adoptive Cell Therapy; Metastatic Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Kidney Neoplasms | interventions — Cyclophosphamide; aldesleukin; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1 (1x10(6) cells (high dose IL-2) (Experimental): Patients will receive (1x10(6) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 2 (3x10(6) cells (high dose IL-2) (Experimental): Patients will receive (3x10(6) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 3 (1x10(7) cells (high dose IL-2) (Experimental): Patients will receive (1x10(7) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 4 (3x10(7) cells (high dose IL-2) (Experimental): Patients will receive (3x10(7) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 5 (1x10(8) cells (high dose IL-2) (Experimental): Patients will receive (1x10(8) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 6 (3x10(8) cells (high dose IL-2) (Experimental): Patients will receive (3x10(8) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 7 (1x10(9) cells (high dose IL-2) (Experimental): Patients will receive (1x10(9) cells plus high dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 8 (1x10(9) cells (low dose IL-2) (Experimental): Patients will receive (1x10(9) cells plus low dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort 9 (3x10(9) cells (low dose IL-2) (Experimental): Patients will receive (3x10(9) cells plus low dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort10(1x10(10) cells (low dose IL-2) (Experimental): Patients will receive (1x10(10) cells plus low dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine
- Cohort11(3x10(10) cells (low dose IL-2) (Experimental): Patients will receive (3x10(10) cells plus low dose aldesleukin
  Interventions: Biological: Anti-VEGFR2 CAR CD8 plus PBL; Drug: Cyclophosphamide; Biological: Aldesleukin; Drug: Fludarabine

INTERVENTIONS:
Biological: Anti-VEGFR2 CAR CD8 plus PBL — Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose (Arms 1-7) or low dose (Arms 8-11) aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose in 5% water (D5W) with mesna 15 mg/kg/day X 2 days over 1 hr
  Other Names: Cytoxan
Biological: Aldesleukin — Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg (Arms 1-7) or 72,000 IU/kg (Arms 8-11) as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Other Names: Proleukin
Drug: Fludarabine — Fludarabine 25 mg/m(2)/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days
  Other Names: Fludara

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients metastatic cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patient s white blood cells with a retrovirus that has the gene for anti-vascular endothelial growth factor receptor (VEGFR2) incorporated in the retrovirus.

Objectives:

- To determine a safe number of these cells to infuse and to see the safety and effectiveness of cell therapy using anti-VEGFR2 gene modified tumor white blood cells to treat recurrent or relapsed cancer.

Eligibility:

- Individuals greater than or equal to 18 years of age and less than or equal to 70 years of age who have been diagnosed with metastatic cancer that has not responded to or has relapsed after standard treatment.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed
* Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti-VEGFR2 cells. {Leukapheresis is a common procedure which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-VEGFR2 cells and aldesleukin. They will stay in the hospital for about4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains a chimeric T cell receptor (CAR) that recognizes the Vascular Endothelial Growth Factor Receptor 2 (VEGFR2), which can be used to mediate genetic transfer of this CAR with high efficiency (> 50%) without the need to perform any selection. Administration of VEGFR2 CAR transduced cells inhibited tumor growth in several different models in different mouse strains.
* In co-cultures with VEGFR2 expressing cells, anti-VEGFR2 transduced T cells secreted significant amounts of interferon (IFN) gamma with high specificity.

Objectives:

Primary objectives:

* To evaluate the safety of the administration of anti-VEGFR2 CAR engineered cluster of differentiation 8 (CD8)+ peripheral blood lymphocytes in patients receiving a non- myeloablative conditioning regimen, and aldesleukin.
* Determine if the administration of anti-VEGFR2 CAR engineered CD8+ peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer.

Secondary objective:

-Determine the in vivo survival of CAR gene-engineered cells.

Eligibility:

Patients who are 18 years of age or older must have:

* metastatic cancer;
* previously received and have been a non-responder to or recurred after standard care for metastatic disease;

Patients may not have:

-contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5 times 10(9) cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) cells to retroviral vector supernatant containing the VEGFR2 genes.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo CAR gene-transduced CD8+ PBMC plus intravenous (IV) aldesleukin. With approval of amendment C, aldesleukin (based on total body weight) will be administered at a dose of 72,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design. Initially, the protocol will enroll 1 patient in each dose cohort unless that patient experiences a dose limiting toxicity (DLT). Should a single patient experience a dose limiting toxicity due to the cell transfer at a particular dose level, additional patients would be treated at that dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose prior to starting the phase II portion. If a dose limiting toxicity occurs in the first cohort, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, the study will be terminated. If IFN-gamma levels increase substantially (as defined in the protocol) in the patient in a cohort compared to the prior patient, the cohort would be expanded to an n=3 to obtain more data on this phenomenon. If one of these 3 patients experience a DLT, the cohort will be expanded to six patients. Following amendment C, patients will be enrolled in cohorts 8-11, with the non-myeloablative chemotherapy regimen, cells and low dose aldesleukin following a conventional 3+3 design. Once the maximum tolerated dose (MTD) has been determined, the study then would proceed to the phase II portion. Patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic melanoma and renal cancer, and cohort 2 will include patients with other types of metastatic cancer.
* For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* The objective will be to determine if the combination of aldesleukin, lymphocyte depleting chemotherapy, and anti-VEGFR2 CAR-gene engineered CD8+ lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic cancer with evaluable disease.
  2. Patients must have previously received at least one systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
  3. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
  4. Willing to sign a durable power of attorney
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
  9. Serology:

     1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
  10. Hematology:

      1. Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim.
      2. White blood cell (WBC) (> 3000/mm(3)).
      3. Platelet count greater than 100,000/mm(3).
      4. Hemoglobin greater than 8.0 g/dl.
  11. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilberts Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
  13. More than 4 weeks must have elapsed since an surgical procedure at the time the patient receives the preparative regimen due to the inhibition of wound healing observed with vascular endothelial growth factor receptor (VEGFR) targeting angiogenesis inhibitors.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Patients with known brain metastases.
3. Patients receiving full dose anticoagulative therapy.
4. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
6. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
7. Patients with diabetic retinopathy.
8. Concurrent Systemic steroid therapy.
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
10. History of coronary revascularization or ischemic symptoms.
11. In patients

Documented forced expiratory volume 1 (FEV1) less than or equal to 45% predicted tested in patients with:

1. History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.
2. Age greater than or equal to 60 years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg SA. Progress in human tumour immunology and immunotherapy. Nature. 2001 May 17;411(6835):380-4. doi: 10.1038/35077246. PMID 11357146
- [Background] Berendt MJ, North RJ. T-cell-mediated suppression of anti-tumor immunity. An explanation for progressive growth of an immunogenic tumor. J Exp Med. 1980 Jan 1;151(1):69-80. doi: 10.1084/jem.151.1.69. PMID 6444236
- [Background] Gattinoni L, Powell DJ Jr, Rosenberg SA, Restifo NP. Adoptive immunotherapy for cancer: building on success. Nat Rev Immunol. 2006 May;6(5):383-93. doi: 10.1038/nri1842. PMID 16622476
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0013.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-four participants were enrolled but one participant was not treated due to a new cancer diagnosis which made the participant ineligible for this protocol.
Groups:
- Cohort 1 - 1 x 10(6) Cells (High Dose IL-2): Anti-vascular endothelial growth factor receptor 2 (VEGFR2) chimeric T cell receptor (CAR) cluster of differentiation 8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 2 - 3 x 10(6) Cells (High Dose IL-2); Cohort 3 - 1 x 10(7) Cells (High Dose IL-2); Cohort 4 - 3 x 10(7) Cells (High Dose IL-2); Cohort 5 - 1 x 10(8) Cells (High Dose IL-2); Cohort 6 - 3 x 10(8) Cells (High Dose IL-2); Cohort 7 - 1 x 10(9) Cells (High Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 8 - 1 x 10(9) Cells (Low Dose IL-2); Cohort 9 - 3 x 10(9) Cells (Low Dose IL-2); Cohort 10 - 1 x 10(10) Cells (Low Dose IL-2); Cohort 11 - 3 x 10(10) Cells (Low Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and low dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 72,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
Period: Overall Study
Arm/Group | Cohort 1 - 1 x 10(6) Cells (High Dose IL-2) | Cohort 2 - 3 x 10(6) Cells (High Dose IL-2) | Cohort 3 - 1 x 10(7) Cells (High Dose IL-2) | Cohort 4 - 3 x 10(7) Cells (High Dose IL-2) | Cohort 5 - 1 x 10(8) Cells (High Dose IL-2) | Cohort 6 - 3 x 10(8) Cells (High Dose IL-2) | Cohort 7 - 1 x 10(9) Cells (High Dose IL-2) | Cohort 8 - 1 x 10(9) Cells (Low Dose IL-2) | Cohort 9 - 3 x 10(9) Cells (Low Dose IL-2) | Cohort 10 - 1 x 10(10) Cells (Low Dose IL-2) | Cohort 11 - 3 x 10(10) Cells (Low Dose IL-2)
Started | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 2
Completed | 1 | 1 | 3 | 1 | 1 | 1 | 3 | 3 | 3 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death during treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - 1 x 10(6) Cells (High Dose IL-2): Anti-vascular endothelial growth factor receptor 2 (VEGFR2) Chimeric T cell receptor (CAR) CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 1 x 10(6) Cells (High Dose IL-2) | Cohort 2 - 3 x 10(6) Cells (High Dose IL-2) | Cohort 3 - 1 x 10(7) Cells (High Dose IL-2) | Cohort 4 - 3 x 10(7) Cells (High Dose IL-2) | Cohort 5 - 1 x 10(8) Cells (High Dose IL-2) | Cohort 6 - 3 x 10(8) Cells (High Dose IL-2) | Cohort 7 - 1 x 10(9) Cells (High Dose IL-2) | Cohort 8 - 1 x 10(9) Cells (Low Dose IL-2) | Cohort 9 - 3 x 10(9) Cells (Low Dose IL-2) | Cohort 10 - 1 x 10(10) Cells (Low Dose IL-2) | Cohort 11 - 3 x 10(10) Cells (Low Dose IL-2) | Total
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 2 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 0 | 1 | 1 | 4 | 3 | 3 | 4 | 2 | 23
  >=65 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (0) | 51.0 (0) | 52.7 (12.1) | 65.0 (0) | 55.0 (0) | 35.0 (0) | 45.5 (11.3) | 37.0 (18.0) | 54.7 (11.9) | 46.3 (5.6) | 41.5 (10.6) | 47.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 7
  Male | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 2 | 2 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 3 | 1 | 1 | 0 | 4 | 3 | 2 | 4 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 3 | 1 | 1 | 0 | 3 | 2 | 3 | 4 | 1 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response to Therapy
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment starts or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - 1x10(6) Cells (High Dose IL-2): Anti-vascular endothelial growth factor receptor 2 (VEGFR2) Chimeric T cell receptor (CAR) CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 2 - 3x10(6) Cells (High Dose IL-2); Cohort 3 - 1x10(7) Cells (High Dose IL-2); Cohort 4 - 3x10(7) Cells (High Dose IL-2); Cohort 5 - 1x10(8) Cells (High Dose IL-2); Cohort 6 - 3x10(8) Cells (High Dose IL-2); Cohort 7 - 1x10(9) Cells (High Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 8 - 1x10(9) Cells (Low Dose IL-2); Cohort 9 - 3x10(9) Cells (Low Dose IL-2); Cohort 10 - 1x10(10) Cells (Low Dose IL-2); Cohort 11 - 3x10(10) Cells (Low Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and low dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 72,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
Arm/Group | Cohort 1 - 1x10(6) Cells (High Dose IL-2) | Cohort 2 - 3x10(6) Cells (High Dose IL-2) | Cohort 3 - 1x10(7) Cells (High Dose IL-2) | Cohort 4 - 3x10(7) Cells (High Dose IL-2) | Cohort 5 - 1x10(8) Cells (High Dose IL-2) | Cohort 6 - 3x10(8) Cells (High Dose IL-2) | Cohort 7 - 1x10(9) Cells (High Dose IL-2) | Cohort 8 - 1x10(9) Cells (Low Dose IL-2) | Cohort 9 - 3x10(9) Cells (Low Dose IL-2) | Cohort 10 - 1x10(10) Cells (Low Dose IL-2) | Cohort 11 - 3x10(10) Cells (Low Dose IL-2)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 2
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Progressive Disease (PD) | 1 | 1 | 3 | 1 | 1 | 1 | 3 | 3 | 3 | 3 | 2
  Stable Disease (SD) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 33 months and 25 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - 1 x 10(6) Cells (High Dose IL-2): Anti-vascular endothelial growth factor receptor 2(VEGFR2) chimeric T cell receptor (CAR) CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
Arm/Group | Cohort 1 - 1 x 10(6) Cells (High Dose IL-2) | Cohort 2 - 3 x 10(6) Cells (High Dose IL-2) | Cohort 3 - 1 x 10(7) Cells (High Dose IL-2) | Cohort 4 - 3 x 10(7) Cells (High Dose IL-2) | Cohort 5 - 1 x 10(8) Cells (High Dose IL-2) | Cohort 6 - 3 x 10(8) Cells (High Dose IL-2) | Cohort 7 - 1 x 10(9) Cells (High Dose IL-2) | Cohort 8 - 1 x 10(9) Cells (Low Dose IL-2) | Cohort 9 - 3 x 10(9) Cells (Low Dose IL-2) | Cohort 10 - 1 x 10(10) Cells (Low Dose IL-2) | Cohort 11 - 3 x 10(10) Cells (Low Dose IL-2)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 2
Participants | 1 | 1 | 3 | 1 | 1 | 1 | 4 | 3 | 3 | 3 | 2

3. Secondary Outcome: In Vivo Survival of Chimeric T Cell Receptor (CAR) Gene-engineered Cells
Description: Immunological monitoring using both tetramer analysis and staining for the T cell receptor (TCR) will be used to augment polymerase chain reaction (PCR)-based analysis. This will provide data to estimate the in vivo survival of lymphocytes derived from the infused cells.
Time Frame: 6 years
Population: This outcome measure was not done due to the lack of a minimum number (e.g. 4) of required durable responses in the participants. A durable response is defined as a complete response, partial response, or stable disease in at least 4 participants.
Arm/Group | Cohort 1 - 1 x 10(6) Cells (High Dose IL-2) | Cohort 2 - 3 x 10(6) Cells (High Dose IL-2) | Cohort 3 - 1 x 10(7) Cells (High Dose IL-2) | Cohort 4 - 3 x 10(7) Cells (High Dose IL-2) | Cohort 5 - 1 x 10(8) Cells (High Dose IL-2) | Cohort 6 - 3 x 10(8) Cells (High Dose IL-2) | Cohort 7 - 1 x 10(9) Cells (High Dose IL-2) | Cohort 8 - 1 x 10(9) Cells (Low Dose IL-2) | Cohort 9 - 3 x 10(9) Cells (Low Dose IL-2) | Cohort 10 - 1 x 10(10) Cells (Low Dose IL-2) | Cohort 11 - 3 x 10(10) Cells (Low Dose IL-2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 33 months and 25 days
Groups:
- Cohort 1 (1x10(6) Cells (High Dose IL-2): Anti-vascular endothelial growth factor receptor 2 (VEGFR2) chimeric T cell receptor (CAR) CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 2 (3x10(6) Cells (High Dose IL-2); Cohort 3 (1x10(7) Cells (High Dose IL-2); Cohort 4 (3x10(7) Cells (High Dose IL-2); Cohort 5 (1x10(8) Cells (High Dose IL-2); Cohort 6 (1x10(8) Cells (High Dose IL-2); Cohort 7 (1x10(9) Cells (High Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and high dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 720,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
- Cohort 8 (1x10(9) Cells (Low Dose IL-2); Cohort 9 (3x10(9) Cells (Low Dose IL-2); Cohort 10 (1x10(10) Cells (Low Dose IL-2); Cohort 11 (3x10(10) Cells (Low Dose IL-2): Anti-VEGFR2 CAR CD8 plus PBL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of anti-VEGFR CAR CD8+ PBL and low dose aldesleukin. On day 0, cells will be infused in the Patient Care Unit over 20-30 minutes (Phase 1: 10e6- 3x10e10 cells and Phase 2: maximum tolerated dose of cells from Phase 1)
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day X 2 days over 1 hr
  Aldesleukin: Aldesleukin (based on total body weight) will be administered at a dose of 72,000 IU/kg as an intravenous bolus over a 15 minute period approximately every eight hours (+/- 1 hour) beginning within 24 hours of the cell infusion and continuing for up to 5 days (maximum 15 doses)
  Fludarabine: Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days
Arm/Group | Cohort 1 (1x10(6) Cells (High Dose IL-2) | Cohort 2 (3x10(6) Cells (High Dose IL-2) | Cohort 3 (1x10(7) Cells (High Dose IL-2) | Cohort 4 (3x10(7) Cells (High Dose IL-2) | Cohort 5 (1x10(8) Cells (High Dose IL-2) | Cohort 6 (1x10(8) Cells (High Dose IL-2) | Cohort 7 (1x10(9) Cells (High Dose IL-2) | Cohort 8 (1x10(9) Cells (Low Dose IL-2) | Cohort 9 (3x10(9) Cells (Low Dose IL-2) | Cohort 10 (1x10(10) Cells (Low Dose IL-2) | Cohort 11 (3x10(10) Cells (Low Dose IL-2)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/1 | 0/1 | 0/1 | 1/4 | 0/3 | 0/3 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/3 | 0/1 | 1/1 | 0/1 | 3/4 | 0/3 | 0/3 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 1/1 | 1/1 | 1/1 | 4/4 | 3/3 | 3/3 | 3/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (1x10(6) Cells (High Dose IL-2) (N=1) | Cohort 2 (3x10(6) Cells (High Dose IL-2) (N=1) | Cohort 3 (1x10(7) Cells (High Dose IL-2) (N=3) | Cohort 4 (3x10(7) Cells (High Dose IL-2) (N=1) | Cohort 5 (1x10(8) Cells (High Dose IL-2) (N=1) | Cohort 6 (1x10(8) Cells (High Dose IL-2) (N=1) | Cohort 7 (1x10(9) Cells (High Dose IL-2) (N=4) | Cohort 8 (1x10(9) Cells (Low Dose IL-2) (N=3) | Cohort 9 (3x10(9) Cells (Low Dose IL-2) (N=3) | Cohort 10 (1x10(10) Cells (Low Dose IL-2) (N=4) | Cohort 11 (3x10(10) Cells (Low Dose IL-2) (N=2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (1x10(6) Cells (High Dose IL-2) (N=1) | Cohort 2 (3x10(6) Cells (High Dose IL-2) (N=1) | Cohort 3 (1x10(7) Cells (High Dose IL-2) (N=3) | Cohort 4 (3x10(7) Cells (High Dose IL-2) (N=1) | Cohort 5 (1x10(8) Cells (High Dose IL-2) (N=1) | Cohort 6 (1x10(8) Cells (High Dose IL-2) (N=1) | Cohort 7 (1x10(9) Cells (High Dose IL-2) (N=4) | Cohort 8 (1x10(9) Cells (Low Dose IL-2) (N=3) | Cohort 9 (3x10(9) Cells (Low Dose IL-2) (N=3) | Cohort 10 (1x10(10) Cells (Low Dose IL-2) (N=4) | Cohort 11 (3x10(10) Cells (Low Dose IL-2) (N=2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Leukocytes (Total WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
PTT (Partial Thromboplstin Time) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual-Other (vision changes) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syndromes - Other (hemaphogocytic syndrome) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (low urine output) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT01218867/Prot_SAP_000.pdf
  • Informed Consent Form (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT01218867/ICF_001.pdf